CLINICAL TRIAL: NCT06472804
Title: Insomnia in Patients With Metastatic Non Small Cell Lung Cancer
Brief Title: Insomnia in Patients With Metastatic Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 19-001466; NCI-2024-04893 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-001466 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo medical chart review and complete a questionnaire on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates how common insomnia (difficulties with sleep) is in patients with lung cancer that has spread from where it first started (primary site) to other places in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the frequency of insomnia in patients with metastatic non-small cell lung cancer.

OUTLINE: This is an observational study.

Patients undergo medical chart review and complete a questionnaire on study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of metastatic non small cell lung cancer

  * Undergoing 1st, 2nd or 3rd line of treatment or are in maintenance therapy
  * Older than 18 years old at the time of diagnosis

Exclusion Criteria:

* Subjects will be excluded if they are considered to have advanced terminal cancer, severe depression or other psychiatric disorder or a sleep disorder other than insomnia (sleep apnea, restless leg syndrome, sleep related disorder of breathing), regular use of psychotropic medication other than hypnotics (eg antidepressants) per chart review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic non small cell lung cancer recruited from Mayo Clinic Oncology Center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of clinically significant insomnia | Baseline
  Will be assessed using the Insomnia Severity Index questionnaire (ISI), is a 7-item self-report questionnaire used to gauge the perceived severity of difficulties initiating sleep, staying asleep, and early morning awakenings, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. ISI score of 15 or greater will be used to categorize clinical insomnia. 0 - 7: no clinically significant insomnia, 8 - 14: subthreshold insomnia, 15 - 21: clinical insomnia (moderate severity), 22 - 28: clinical insomnia (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Leventakos, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials